CLINICAL TRIAL: NCT02584946
Title: Effect of Avenanthramides Supplement on Exercise-induced Physiological and Psychological Changes
Brief Title: Avenanthramides and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1513
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Avenanthramides
MeSH Terms: interventions — avenanthramide-2C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-AVA oat flour cookies (Placebo Comparator)
  Interventions: Other: Avenanthramides
- High-AVA oat flour cookies (Experimental)
  Interventions: Other: Avenanthramides

INTERVENTIONS:
Other: Avenanthramides — AVAs are a group of diphenolic acids that are found only in oats (Avena sativa).

SUMMARY:
The aim of the proposed study is to examine whether long-term dietary supplementation (8 weeks) of an oat flour cookie rich in avenanthramides (AVA) could enhance blood antioxidant capacity and reduce blood inflammatory markers after a downhill running (DR) protocol among human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female non-obese subjects (18kg/M2<BMI<28kg/M2) (age 20-45 years) will be recruited from the Twin Cities community. All participants will sign informed consent approved by UMN-IRB and are willing to avoid oat consumption and rigorous physical activity the day prior to and through test and to consume a low-polyphenol diet for 1 week prior to the study. The foods rich in polyphenols include all berries, apples, pears, citrus fruits, fruit juices, onions, chocolate, wine, coffee, tea, beans, nuts, soy products and most spices

Exclusion Criteria:

1. Presence of GI conditions that interfere with absorption;
2. Clinically significant endocrine, cardiovascular, pulmonary, renal, hepatic, pancreatic, biliary or neurologic disorders;
3. Major trauma or surgery within 3 months of visit;
4. Cancer in the prior 2 years;
5. Allergic to oat products;
6. Women who are pregnant or lactating;
7. Smoking;
8. Drinking alcohol >5 drinks/week;
9. Using nutraceuticals;
10. Blood pressure medication;
11. NSAID (>800 mg ibuprofen/week)
12. Vitamin supplementation
13. Anticoagulants or hypoglycemic drugs
14. Oat products consumption and rigorous physical activity the day before the test and consumption of a high-polyphenol diet in week prior to the test.
15. Moderate-intensity cardiorespiratory exercise training for ≥30 min•d-1 on ≥5 d•wk-1 for a total of ≥150 min•wk-1, vigorous-intensity cardiorespiratory exercise training for ≥20 min•d-1 on ≥3 d•wk-1 (≥75 min•wk-1), or a combination of moderate- and vigorous-intensity exercise to achieve a total energy expenditure of ≥500-1000 MET•min•wk-1

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
Mean and SD of plasma concentrations of Creatine Kinase | 0-72 hours

SECONDARY OUTCOMES:
Mean and SD of plasma concentrations of TNF-α | 0-72 hours
Mean and SD of plasma concentrations of IL-6 | 0-72 hours
Mean and SD of plasma concentrations of ICAM-1, VCAM-1, NF-κB (P65), NRB, NF-κB binding to DNA, 4-Hydroxynenenol, F2-isoprostane | 0-72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Li Li Ji, PhD, Principal Investigator — University of Minnesota

REFERENCES:
- [Derived] Zhang T, Zhao T, Zhang Y, Liu T, Gagnon G, Ebrahim J, Johnson J, Chu YF, Ji LL. Avenanthramide supplementation reduces eccentric exercise-induced inflammation in young men and women. J Int Soc Sports Nutr. 2020 Jul 25;17(1):41. doi: 10.1186/s12970-020-00368-3. PMID 32711519